CLINICAL TRIAL: NCT00286286
Title: Clinical Protocol for the Prospective Double Blind Randomised Controlled Trial for the Use of Intraperitoneal Aerosolized Local Anesthetic
Brief Title: Intraperitoneal Aerosolized Delivery of a Local Anesthetic for Post Operative Pain Management. A Double Blind, Randomised Controlled Clinical Trial.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Northgate Technologies (Industry)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: ABHN0635
Record Dates: First submitted 2006-02-01; First posted 2006-02-03 (Estimated); Last update posted 2007-01-11 (Estimated); Status verified 2007-01

CONDITIONS: Pain, Postoperative; Postoperative Pain; Abdominal Pain; Obesity; Pneumoperitoneum
Keywords: Laparoscopy; Laparoscopic Surgical Procedures; Laparoscopic Surgery; Gastric Bypass; Drug Delivery Systems; Pain Measurement
MeSH Terms: conditions — Pain, Postoperative; Abdominal Pain; Obesity; Pneumoperitoneum

INTERVENTIONS:
Device: Intraperitoneal Aerosolization System, IntraMyst

SUMMARY:
The purpose of this study is to determine the effectiveness of aerosolized pain medication (.5% bupivicaine) delivered into the peritoneal cavity after laparoscopic gastric bypass surgery. This double blind study will include 50 patients. 25 will receive the aerosolized pain medication and 25 will receive a placebo (normal saline). All 50 patients will receive routine/typical methods of post-operative pain management. Post operative pain scores of the patients will be examined to determine the effect of aerosolization.

DETAILED DESCRIPTION:
Surgical Technique

1. 30 mls of 0.5% bupivacaine with epinephrine standard dose will be distributed into the trocar site wounds after desufflation of the peritoneal cavity.
2. All the patients will be under a consistent intra-abdominal pressure using CO2 and the laparoscopy will be carried out using the same, routine / typical surgical instruments.

A. Control Group (n=25): Aerosolized normal saline will be introduced at the end of the procedure, using a specially designed sterile catheter. The catheter will be inserted via trocar port under direct vision. The other end of the catheter will be connected to a 72" Edwards Lifesciences pressure tubing (Ref: 50P172), which will be connected to a B&D 20cc syringe filled with 15 ml of normal saline and inserted into a specially designed syringe pump and pressurizing system designed to aerosolize the specified agent. The total dose of patient delivered normal saline will be 10 ml, with 5 ml remaining contained and undelivered within the catheter and 72" pressure tubing. Routine/Typical methods of post-operative pain management will be employed.

B. Aerosolized anesthetic (n=25): at the end of the procedure, the aerosolized local anesthetic will be introduced using a specially designed sterile catheter. The catheter will be inserted via trocar port under direct vision. The other end of the catheter will be connected to a 72" Edwards Lifesciences pressure tubing (Ref: 50P172), which will be connected to a B&D 20cc syringe filled with 15 ml of anesthetic agent and inserted into a specially designed syringe pump and pressurizing system designed to aerosolize the specified agent. The total dose of patient delivered anesthetic will be 10 ml, with 5 ml remaining contained and undelivered within the catheter and 72" pressure tubing. Routine/Typical methods of post-operative pain management will be employed.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients between the ages of 18-65
2. Patients in general good health requiring elective surgery

Exclusion Criteria:

1. Female patients that are pregnant
2. Patients allergic to bupivicaine
3. Patients who have used narcotic drugs within 30 days of the surgical procedure.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2006-02; Study Completion 2006-08

PRIMARY OUTCOMES:
Baseline Pain score before surgery
First Pain score upon arrival in PACU
6 hrs after first recorded pain score
12 hrs after first recorded pain score
24 hrs after first recorded pain score

CONTACTS AND LOCATIONS:
Overall Officials: Peter C. Rantis Jr., MD, Principal Investigator — Alexian Brothers Hospital Network
Locations (2):
- United States (2):
  - Alexian Brothers Medical Center, Elk Grove Village, Illinois
  - St. Alexius Medical Center, Hoffman Estates, Illinois